CLINICAL TRIAL: NCT05283538
Title: Comparison of Cardiovascular Risk Stratification in Young People With Type 1 Diabetes by Coronary Calcium Score to ESC/ESA2019 Recommendations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CACD1
Record Dates: First submitted 2022-01-04; First posted 2022-03-17 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Type 1 Diabetes; Coronary Artery Calcification
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Coronary Artery Calcification Evaluation (Experimental)
  Interventions: Diagnostic Test: Coronary Artery Calcification Realization

INTERVENTIONS:
Diagnostic Test: Coronary Artery Calcification Realization — Coronary Artery Calcification Realization

SUMMARY:
The aim of the study is to compare ESC recommendations on cardiovascular (CV) risk stratification with the achievement of a CAC (Coronary Artery Calcification).

The development of a CAC, currently not systematically offered to these patients to refine CV risk, could make it possible to offer more intensive management of CV risk facors for patients who objectively have a high CV risk as evidenced by a high coronary calcium score.

LDL target recommandations have become more aggressive with a very high level of evidence in type 2 diabetic patients but low in type 1 diabetic patients because there is no specific CV intervention study for T1D patients.

These recommendations have far-reaching consequences because they would justify introducing in young type 1 diabetic patients, considered from the outset to be at moderate cardiovascular risk (young T1DM <35 years old) or even at high cardiovascular risk (duration of diabetes > 10 years) or very high cardiovascular risk (duration of diabetes > 20 years), treatment with statins or even aspirin, based only on the length of time they have had diabetes.

The realization of a CAC, currently not systematically offered to these patients to refine CV risk, could make it possible to propose a more intensive management of CV risk factors for patients with objectively high CV risk attested by a high coronary calcium score.

In this case the introduction of treatment with statins would be indicated.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years and ≤ 35 years; Type 1 diabetic patient (defined by T1DM antibody positivity or onset in pediatric age); In primary cardiovascular prevention (with no CV events); Patient not treated by statins; Duration of diabetes > 5 years; Equipped with a continuous interstitial glucose measurement system for at least 14 days; No previous CAC performed Patient with social security or with third party coverage. Free subject, without guardianship or curatorship or subordination; Informed consent signed by the patient after clear and fair information about the study.

Exclusion Criteria:

* Cardiovascular secondary prevention patients (with a previous CV event); ECG abnormality suggestive of coronary ischemia; Intolerance or contraindication to statins Person benefiting from reinforced protection, namely minors, persons deprived of their liberty by a judicial or administrative decision, persons staying in a health or social establishment, adults under legal protection and finally patients in emergency situations; Pregnant and/or breastfeeding woman.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Statin prescription indication based on the patient's LDL cholesterol value and the LDL cholesterol target determined according to the cardiovascular risk level calculated with the coronary calcium score | 1 day
  The prescription indication is LDL-cholesterol levels above the target level defined according to the level of cardiovascular risk: Moderate< 1 g/l- High< 0.7g/l-Very high< 0.55 g/l
  Coronary calcium score classified according to a consensus of the French Society of Cardiology and the French speaking Society of Diabetology 2020 : Moderate CAC ≤ 10- High 11 ≤ CAC ≤ 100- Very high CAC >100
Statin prescription indication based on the patient's LDL cholesterol value and the LDL cholesterol target determined according to the cardiovascular risk level according to the ESC/ESA 2019 recommendations | 1 day
  The prescription indication is LDL-cholesterol levels above the target level defined according to the level of cardiovascular risk: Moderate< 1 g/l- High< 0.7g/l-Very high< 0.55 g/l
  ESC/ESA 2019 LDL target recommendations are cited in the summary

CONTACTS AND LOCATIONS:
Locations (1):
- C.H.U. de Poitiers, Poitiers, France